CLINICAL TRIAL: NCT04007653
Title: Long-term Outcome After Edoxaban Versus Vitamin K Antagonists for Acute VTE
Acronym: HOKUSAIpostVTE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, S. Middeldorp, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: HOKUSAI post VTE study
Record Dates: First submitted 2019-07-01; First posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Venous Thromboembolic Disease; Post Thrombotic Syndrome; Chronic Thromboembolic Pulmonary Hypertension; Quality of Life
Keywords: Post thrombotic syndrome; Edoxaban; Vitamin K antagonist; Chronic Thromboembolic Pulmonary Hypertension; Quality of Life
MeSH Terms: conditions — Postthrombotic Syndrome | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients treated with heparin+edoxaban for VTE: Patients treated with heparin+edoxaban for a venous thromboembolic event during the HOKUSAI trial, for which they were randomised.
  Interventions: Other: Observation
- Patients treated with heparin+VKA for VTE: Patients treated with heparin+VKA for a venous thromboembolic event during the HOKUSAI trial, for which they were randomised.
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — No intervention

SUMMARY:
The HOKUSAI post VTE study contains of two different research questions; one on the long term outcomes of deep vein thrombosis and one on the long term effects of pulmonary embolism, post thrombotic syndrome (PTS) and chronic thromboembolic pulmonary hypertension (CTEPH) respectively. Our aim of the study is to compare the long term outcomes along with the quality of life assessment of VTE in a group treated with heparin+VKA versus a group treated with heparin+edoxaban in the acute setting.

ELIGIBILITY:
Inclusion Criteria:

* Participant in the HOKUSAI VTE trial

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who were included in the HOKUSAI VTE trial for treatment of their DVT or PE.
Sampling Method: Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2017-04-25 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Post thrombotic syndrome (PTS) | up to 10 years
  PTS according to Villalta

SECONDARY OUTCOMES:
Chronic thromboembolic pulmonary hypertension (CTEPH) | up to 10 years
  according to clinical and objective criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Academisch Medisch Centrum, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided